CLINICAL TRIAL: NCT02829528
Title: Little Flower Yoga for Kids: Evaluation of a Yoga and Mindfulness Program for Children With Increased Levels of Emotion Dysregulation and Inattention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Little Flower Yoga for Kids
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2018-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Little Flower Yoga For Kids (Experimental): Little Flower Yoga for Kids is a New York based organization dedicated to making the tools of yoga and mindfulness available to all children and teens. Their Teacher Training Program focuses on the physical, mental emotional, and social wellbeing of students. Teachers are trained to use the five elements format (connect, breathe, move, focus, relax). Implementation of the Little Flower Yoga for Kids curriculum will be manualized prior to the start of the study with Ms. Love, and will be presented as a series of activities (e.g., poses) throughout the school year. The emphasis in these yoga and mindfulness activities is exploration not competition, which allows the child to learn and develop at her own pace with the support of Ms. Love. The children participate in the Little Flower Yoga for Kids intervention at school for 40 minutes per class, 3 to 5 times per week, for the entire academic school year (9 months).
  Interventions: Behavioral: Little Flower Yoga For Kids

INTERVENTIONS:
Behavioral: Little Flower Yoga For Kids — Little Flower Yoga for Kids is a promising yoga and mindfulness program for children developed by Jennifer Cohen Harper, MA, E-RCYT, which incorporates five elements (connect, breathe, move, focus, relax) to improve the child's ability to sustain attention and regulate emotions.

SUMMARY:
An initial evaluation of Little Flower Yoga for Kids will be conducted in a small sample of 18-30 Kindergarten and First Grade students (3-5 per class) enrolled in Girls Preparatory Charter School of the Bronx. The overall aim of this study is to ascertain the short and longer-term effects of Little Flower Yoga for Kids, a promising yoga and mindfulness program for children, which incorporates five elements (connect, breathe, move, focus, relax) to improve the child's ability to sustain attention and regulate emotions.

DETAILED DESCRIPTION:
The overall aim of this project is to ascertain the effects of Little Flower Yoga for Kids, a promising yoga and mindfulness program for children developed by Jennifer Cohen Harper, MA, E-RCYT, which incorporates five elements (connect, breathe, move, focus, relax) to improve the child's ability to sustain attention and regulate emotions. While research supports that yoga programs and mindfulness programs yield positive outcomes on numerous factors, there are no independent studies presently examining the effects of a combined yoga and mindfulness intervention (like Little Flower Yoga for Kids) on both emotion regulation and sustained attention.

The investigators propose conducting an initial evaluation of Little Flower Yoga for Kids in a small sample of 18-30 Kindergarten and First Grade students (3-5 per class) enrolled in Girls Preparatory Charter School of the Bronx. Little Flower Yoga for Kids is currently part of the curriculum at Girls Preparatory Charter School of the Bronx and implemented by Kelli Love, M.Ed., 500 RYT, received her certification from the Little Flower Yoga for Kids Teacher Training Program. Specifically, the investigators will conduct a preliminary trial with a sample of 5-7 year olds (Kindergarten/First Grade), who meet a predetermined threshold of having either emotional regulation and/or attentional difficulties, to determine the effects of Little Flower Yoga for Kids on sustained attention and emotion regulation. Measures of these outcomes will occur at initial participant screener, baseline, mid-treatment (4.5 months after the start of the program), and post-treatment (after 9 months).

ELIGIBILITY:
While all students enrolled in kindergarten or first grade at Girls Preparatory Charter School of the Bronx (between the ages of 5-7) will continue to take yoga class (with the Little Flower Yoga program Curriculum) taught by Ms. Keli Love, the investigators will only be collecting data on (at most) 30 of the students. The following inclusion and exclusion criteria will be employed to determine which students will be included in the data collection:

Inclusion Criteria:

* Suspected emotion regulation and/or attention difficulties by the child's teacher. This procedure includes completion (by the teacher) of the Emotion Regulation Checklist (ERC) and the inattention subscale of the Swanson, Nolan, and Pelham - IV (SNAP-IV) (see measures section below). The Kindergarten and First Grade teachers will be asked to identify the top 5 students in their class exhibiting high levels of emotion dysregulation and/or inattention in comparison to their peers, and to then fill out the two assessment measures for each of the 5 selected children. They must meet a predetermined threshold of either measure, which have been determined based on previous research, to be included in the data collection;
* Child must be fluent English speaker, so they are able to complete the assessments.

Exclusion Criteria:

Of the individuals chosen for participation in data collection, they will be excluded from the study if:

* There is evidence of significant developmental delay or psychosis that impacts the child's ability to function and to fully engage in the yoga-mindfulness intervention;
* If the youth or parent presents with emergency psychiatric needs that require services beyond that which can be managed within a preventive intervention format (e.g. hospitalization, specialized placement outside the home), active intervention by research staff to secure what is needed will be made.

Ages: 5 Years to 7 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation Content Scale of the Behavioral Assessment System for Children - 2 (BASC-2) | Nine months from start of the intervention
  Measures change in emotion regulation problems at post-treatment
Tasks of Executive Control (TEC) | Nine months from start of the intervention
  Measures change in attentional processing skills at post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

REFERENCES:
- See also: Description: Families and Children Experiencing Success (FACES) Lab — http://steinhardt.nyu.edu/appsych/faceslab